CLINICAL TRIAL: NCT06519422
Title: The Effects of Tranexamic Acid on Anaemia, Menstrual Health and the Wellbeing of Women: an International Randomised, Placebo-controlled Trial Among Menstruating Women With Anaemia
Brief Title: Tranexamic Acid for Anaemia Trial
Acronym: WOMAN-3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: The Jon Moulton Charity Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WOMAN-3
Record Dates: First submitted 2024-07-11; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Anemia
Keywords: Tranexamic acid; Antifibrinolytic; Anaemia; Menstrual health; Menstruation; Bleeding
MeSH Terms: conditions — Anemia; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (TXA) (Experimental): Tranexamic acid 1 gram (2x 500 mg) orally taken three times a day from the first to the last day of the menstrual period for up to 5 days, for 3 successive periods.
  Interventions: Drug: Tranexamic Acid 500 MG
- Placebo (Placebo Comparator): Matched placebo tablets taken three times a day from the first to the last day of the menstrual period for up to 5 days, for 3 successive periods.
  Interventions: Other: Matched placebo

INTERVENTIONS:
Drug: Tranexamic Acid 500 MG — Tablets
  Arms: Tranexamic acid (TXA)
Other: Matched placebo — Matched placebo tablets (inactive ingredients only, including microcrystalline cellulose, magnesium stearate BP and lactose)
  Arms: Placebo

SUMMARY:
Anaemia is a common health problem in women. It is often due to iron deficiency. Anaemia is a particular problem during pregnancy and is bad for the mother and baby. It is best to treat anaemia in young women well before they get pregnant. Doctors treat anaemia with iron and vitamins. But some people get side effects when taking iron tablets and so they stop taking them. Heavy menstrual periods are a common cause of iron deficiency and even if women do take iron, because they lose so much iron in their periods, they still become iron deficient. Tranexamic acid (TXA) is a medicine used to treat heavy periods. The investigators of this study would like to find out if taking TXA with the usual iron and vitamin supplements is better at treating anaemia than taking iron and vitamin supplements alone. (Lay Summary)

DETAILED DESCRIPTION:
World-wide, half a billion women of reproductive age are anaemic. Anaemia has major health consequences for pregnant women and their babies. Anaemia increases the risk of ante-partum haemorrhage, prematurity, stillbirth, neonatal death, post-partum haemorrhage and maternal death. Early intervention to reduce the risk of anaemia before pregnancy offers the potential to reduce adverse maternal and birth outcomes and improve well-being across the reproductive life course.

Unfortunately, global efforts to reduce anaemia prevalence by 2025 are far off track. Anaemia worsens bleeding through multiple biological mechanisms. Anaemia increases blood flow from bleeding vessels due to reduced blood viscosity and anaemic blood clots are more susceptible to fibrinolysis. Although iron and multivitamin replacement is the mainstay of anaemia treatment, iron stores in young women depend more on menstrual iron loss than on dietary intake. Because anaemia worsens bleeding, women with anaemia have heavier menstrual periods than if they were not anaemic. For this reason, offering iron replacement without reducing menstrual iron loss may be inefficient.

The antifibrinolytic tranexamic acid (TXA) reduces menstrual bleeding by preventing blood clot breakdown. The investigators propose that giving TXA with iron and vitamin replacement will be more effective in treating anaemia than iron and vitamin replacement alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (aged 18 years and older)
* Having menstrual periods every 21 to 38 days that last 2 to 9 days
* Having anaemia (Hb < 120 g/L) according to point-of-care finger prick screening test
* Willing to provide informed consent and able to attend study visits during the trial period

(Individuals with known thalassaemia are eligible to participate and take the trial treatment but will not receive standard of care iron supplementation. They will continue to receive their standard care.)

Exclusion Criteria:

* Planning to get pregnant during trial period
* Already taking TXA
* Known to have contraindications to TXA treatment (including allergy to TXA or its excipients, renal impairment, active thromboembolic disease, history of venous or arterial thrombosis, history of convulsion.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Anaemia | After the 3rd and before the 4th menstrual period or by 6 months from baseline, whichever occurs first.
  The proportion of participants with anaemia, defined as Haemoglobin (Hb) < 120 g/L (measured on venous blood)

SECONDARY OUTCOMES:
Haemoglobin (Hb) concentration | After the 3rd and before the 4th menstrual period or by 6 months from baseline, whichever occurs first.
  Hb measured on venous blood
Severity of anaemia | After the 3rd and before the 4th menstrual period or by 6 months from baseline, whichever occurs first.
  Mild Anaemia (Hb=110-119 g/L); Moderate Anaemia (Hb=80-109 g/L); Severe Anaemia (Hb < 80 g/L); Hb measured on venous blood
Ferritin | After the 3rd and before the 4th menstrual period or by 6 months from baseline, whichever occurs first.
  Serum ferritin (from venous blood sample) and CRP-adjusted ferritin (see below, under C-reactive protein)
Iron deficiency | After the 3rd and before the 4th menstrual period or by 6 months from baseline, whichever occurs first.
  Iron deficiency defined as ferritin <15 ug/L (WHO definition) and defined as ferritin <30 ug/L, (new clinical consensus); Serum ferritin from venous blood sample; CRP-adjusted ferritin (see below, under C-reactive protein)
  Note: CRP-adjusted ferritin (see below)
C-reactive protein (CRP) | After the 3rd and before the 4th menstrual period or by 6 months from baseline, whichever occurs first.
  The Statistical Analysis Plan (SAP) will include details on how ferritin values will be corrected by taking into account CRP levels (inflammation marker), because normal ferritin concentrations may mask an iron deficient state if inflammation is present
Iron-deficiency anaemia | After the 3rd and before the 4th menstrual period or by 6 months from baseline, whichever occurs first.
  The proportion of participants with iron-deficiency anaemia, defined as presence of both anaemia (Hb<120 g/L) plus iron deficiency (ferritin <15 ug/L AND/OR <30 ug/L), measured as detailed above (using CRP-adjusted ferritin levels, as explained above)
Menstrual blood loss | During 3 menstrual periods (on average about 3 months, but no longer than 6 months from baseline)
  Blood loss assessed semi-quantitatively by pictorial blood assessment chart (PBAC), adapted from Higham et al (1990), DOI: 10.1111/j.1471-0528.1990.tb16249.x
Perceived change in menstrual blood loss | After the 3rd and before the 4th menstrual period or by 6 months from baseline, whichever occurs first.
  Participant's subjective assessment of change in menstrual bleeding from baseline, e.g. expressed on a Likert scale ('greatly improved' to 'much worse')
Degree of effect of menstrual bleeding on health-related Quality of Life | After the 3rd and before the 4th menstrual period or by 6 months from baseline, whichever occurs first.
  SAMANTA scale (ref: Calaf, 2020, DOI: 10.1089/jwh.2018.7446 and Sinharoy 2023, DOI: 10.1016/S2214-109X(23)00416-3; Affirmative answers to two questions ('experiencing menstrual bleeding for >7 days per month' and 'being bothered by menstruation due to its Abundance') each receive 3 points, while affirmative answers to all other questions each receive 1 point ('≥3 days of heavier bleeding', 'blood spotting on clothes at night', 'worried about staining furniture', 'avoid some activities because of the need to change menstrual materials'). These values are summed, resulting in a potential range of values for the heavy menstrual bleeding score from 0 to 10.)
Flooding | During 3 menstrual periods (on average about 3 months, but no longer than 6 months from baseline)
  'Flooding' experienced during menstrual period (provisionally defined by Cooper 2013, DOI: 10.1111/1471-0528.17473, as "sudden overwhelming blood loss that exceeds the saturation of the menstrual products being used")

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sima Berendes, Study Director — London School of Hygiene and Tropical Medicine (Clinical Trials Unit)

IPD SHARING:
Plan to Share IPD: Yes
We are committed to sharing data for ethical research with justified scientific objectives. Until all planned analyses are completed by the LSHTM CTU Global Health Trials Group, data will be shared through a controlled access approach; thereby researchers can make formal applications for data sharing. Afterwards, we will share the anonymised dataset via the LSHTM CTU Global Health Trials Group data sharing platform at freebird.lshtm.ac.uk or a similar platform. We will make all relevant trial materials available on the trial website.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once all planned analyses are completed by the LSHTM CTU Global Health Trials Group following trial completion. Data will be shared indefinitely.
Access Criteria: As described above
URL: http://freebird.lshtm.ac.uk